CLINICAL TRIAL: NCT02693535
Title: Targeted Agent and Profiling Utilization Registry (TAPUR) Study
Brief Title: TAPUR: Testing the Use of Food and Drug Administration (FDA) Approved Drugs That Target a Specific Abnormality in a Tumor Gene in People With Advanced Stage Cancer
Acronym: TAPUR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American Society of Clinical Oncology (Other)
Collaborators: AstraZeneca (Industry); Bayer (Industry); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry); Genentech, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Boehringer Ingelheim (Industry); Seagen Inc. (Industry); Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014171
Record Dates: First submitted 2016-02-11; First posted 2016-02-26 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma; Advanced Solid Tumors
Keywords: cancer; off-label; precision medicine; targeted therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma; Neoplasms | interventions — palbociclib; Sunitinib; temsirolimus; Trastuzumab; pertuzumab; Vemurafenib; cobimetinib; regorafenib; olaparib; pembrolizumab; Nivolumab; Ipilimumab; abemaciclib; talazoparib; atezolizumab; entrectinib; larotrectinib; tucatinib; futibatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (17):
- Group 4 (CDKN2A, CDK4, CDK6) (Other): Participants receive palbociclib - dosage, frequency and duration per label; acceptable genomic matches include CDKN2A loss or mutation, CDK4, CDK6 amplifications, CDKN2B loss or mutation
  Interventions: Drug: Palbociclib
- Group 5 (CSF1R,PDGFR,VEGFR) (Other): Participants receive sunitinib - dosage, frequency and duration per label; acceptable genomic matches include CSF1R, PDGFR, VEGFR1/2/3, KIT, FLT-3, RET, FGFR1/2/3, VHL amplifications or mutations
  Interventions: Drug: Sunitinib
- Group 6 (mTOR, TSC) (Other): Participants receive temsirolimus - dosage, frequency and duration per label; acceptable genomic matches include mTOR, TSC1/2, AKT1 mutations
  Interventions: Drug: Temsirolimus
- Group 8 (ERBB2) (Other): Participants receive trastuzumab and pertuzumab - dosage, frequency and duration per label; acceptable genomic matches include ERBB2 amplification or overexpression, and specific ERBB2 mutations
  Interventions: Drug: Trastuzumab and Pertuzumab
- Group 9 (BRAF V600E/D/K/R) (Other): Participants receive vemurafenib and cobimetinib - dosage, frequency and duration per label; acceptable genomic matches include BRAF V600E/D/K/R mutations
  Interventions: Drug: Vemurafenib and Cobimetinib
- Group 13 (RET,VEGFR1/2/3,KIT,PDGFRβ,RAF-1,BRAF) (Other): Participants receive regorafenib - dosage, frequency and duration per label; acceptable genomic matches include RET, VEGFR1/2/3, KIT, PDGFRβ, RAF-1, BRAF mutations or amplifications
  Interventions: Drug: Regorafenib
- Group 14 (BRCA1/2; ATM) (Other): Participants receive olaparib - dosage, frequency and duration per label; acceptable genomic matches include germline or somatic BRCA1/2 inactivating mutations; ATM mutations or deletions
  Interventions: Drug: Olaparib
- Group 15 (POLE, POLD1) (Other): Participants receive pembrolizumab - dosage, frequency and duration per label; acceptable genomic matches include specific POLE and POLD1 mutations
  Interventions: Drug: Pembrolizumab
- Group 16 (MSI-H, high mutational load and others) (Other): Participants receive nivolumab and ipilimumab - dosage, frequency and duration per label; acceptable genomic matches include MSI high status, high tumor mutational burden, MLH1, MSH2/6, PMS2, EPCAM mutations, specific POLE or POLD1 mutations, BRCA1/2, ATM, MSH3, PMS1, MLH3, EXO1, RFC1/2/3/4/5, PCNA, RPA1/2/3/4, and SSBP1 loss of function mutations
  Interventions: Drug: Nivolumab and Ipilimumab
- Group 17 (CDKN2A, CDK4, CDK6) (Other): Participants receive abemaciclib - dosage, frequency and duration per label; acceptable genomic matches include CDKN2A loss or mutation, CDK4, CDK6 amplifications, CDKN2B loss or mutation
  Interventions: Drug: Abemaciclib
- Group 19 (BRCA1/2, PALB2) (Other): Participants receive talazoparib - dosage, frequency and duration per label; acceptable genomic matches include germline or somatic BRCA1/2 and PALB2 mutations
  Interventions: Drug: Talazoparib
- Group 20 (ERBB2) (Other): Participants receive atezolizumab plus PHESGO - dosage, frequency and duration per label; acceptable genomic matches include ERBB2 amplification or overexpression
  Interventions: Drug: Atezolizumab and PHESGO
- Group 21 (BRCA1/2, PALB2, ATM, and others) (Other): Participants receive atezolizumab plus talazoparib - dosage, frequency and duration per label; acceptable genomic matches include germline or somatic mutations in BRCA1/2, PALB2, ATM, ATR, CHEK2, FANCA, RAD51C, NBN, MLH1, MRE11A, CDK12; positive genomic instability score reported on the Myriad MyChoice CDx test; or Genomic Loss of Heterozygosity (LOH) Score above threshold as reported on a FoundationOne CDx test or another qualifying test for TAPUR with MTB approval
  Interventions: Drug: Atezolizumab and Talazoparib
- Group 22 (ROS1 fusion) (Other): Participants receive entrectinib - dosage, frequency and duration per label; acceptable genomic matches include any ROS1 fusion
  Interventions: Drug: Entrectinib
- Group 23 (NTRK amplification) (Other): Participants receive larotrectinib - dosage, frequency and duration per label; acceptable genomic matches include NTRK1/2/3 amplification
  Interventions: Drug: Larotrectinib
- Group 24 (ERBB2) (Other): Participants receive tucatinib plus trastuzumab SC - dosage, frequency and duration per label; acceptable genomic matches include ERBB2 amplification or overexpression, and specific ERBB2 mutations
  Interventions: Drug: Tucatinib plus Trastuzumab Subcutaneous (SC)
- Group 25 (Other): Participants receive futibatinib- dosage, frequency and duration per label; acceptable genomic matches include FGFR 1,2,3,4 fusion (or other rearrangement) or mutation
  Interventions: Drug: Futibatinib

INTERVENTIONS:
Drug: Palbociclib — drug
  Other Names: Ibrance
  Arms: Group 4 (CDKN2A, CDK4, CDK6)
Drug: Sunitinib — drug
  Other Names: Sutent
  Arms: Group 5 (CSF1R,PDGFR,VEGFR)
Drug: Temsirolimus — drug
  Other Names: Torisel
  Arms: Group 6 (mTOR, TSC)
Drug: Trastuzumab and Pertuzumab — drug
  Other Names: Herceptin and Perjeta
  Arms: Group 8 (ERBB2)
Drug: Vemurafenib and Cobimetinib — drug
  Other Names: Zelboraf and Cotellic
  Arms: Group 9 (BRAF V600E/D/K/R)
Drug: Regorafenib — drug
  Other Names: Stivarga
  Arms: Group 13 (RET,VEGFR1/2/3,KIT,PDGFRβ,RAF-1,BRAF)
Drug: Olaparib — drug
  Other Names: Lynparza
  Arms: Group 14 (BRCA1/2; ATM)
Drug: Pembrolizumab — drug
  Other Names: Keytruda
  Arms: Group 15 (POLE, POLD1)
Drug: Nivolumab and Ipilimumab — drug
  Other Names: Opdivo and Yervoy
  Arms: Group 16 (MSI-H, high mutational load and others)
Drug: Abemaciclib — drug
  Other Names: Verzenio
  Arms: Group 17 (CDKN2A, CDK4, CDK6)
Drug: Talazoparib — drug
  Other Names: Talzenna
  Arms: Group 19 (BRCA1/2, PALB2)
Drug: Atezolizumab and PHESGO — drug
  Other Names: Tecentriq and PHESGO
  Arms: Group 20 (ERBB2)
Drug: Atezolizumab and Talazoparib — drug
  Other Names: Tecentriq and Talzenna
  Arms: Group 21 (BRCA1/2, PALB2, ATM, and others)
Drug: Entrectinib — drug
  Other Names: Rozlytrek
  Arms: Group 22 (ROS1 fusion)
Drug: Larotrectinib — drug
  Other Names: Vitrakvi
  Arms: Group 23 (NTRK amplification)
Drug: Tucatinib plus Trastuzumab Subcutaneous (SC) — drug
  Other Names: Tukysa and Herceptin Hylecta
  Arms: Group 24 (ERBB2)
Drug: Futibatinib — drug
  Other Names: Lytgobi
  Arms: Group 25

SUMMARY:
The purpose of the study is to learn from the real world practice of prescribing targeted therapies to patients with advanced cancer whose tumor harbors a genomic variant known to be a drug target or to predict sensitivity to a drug.

NOTE: Due to character limits, the arms section does NOT include all TAPUR Study relevant biomarkers. For additional information, contact TAPUR@asco.org, or if a patient, your nearest participating TAPUR site (see participating centers).

********************************************************************

Results in publication or poster presentation format are posted as they become available for individual cohorts at www.tapur.org/news. The results may be accessed at any time. All results will be made available on clinicaltrials.gov at the end of the study. Indexing of available results on PubMed is in progress.

********************************************************************

DETAILED DESCRIPTION:
The Targeted Agent and Profiling Utilization Registry (TAPUR) Study is a non-randomized clinical trial that aims to describe the safety and efficacy of commercially available, targeted anticancer drugs prescribed for treatment of patients with advanced cancer that has a potentially actionable genomic variant. TAPUR will study Food and Drug Administration (FDA)-approved targeted therapies that are contributed by collaborating pharmaceutical companies, catalogue the choice of molecular profiling test by clinical oncologists and develop hypotheses for additional clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older (*Restrictions apply. Not all therapies are available for patients <18)
* Histologically-proven locally advanced or metastatic solid tumor, multiple myeloma or B cell non-Hodgkin lymphoma who is no longer benefiting from standard anti-cancer treatment or for whom, in the opinion of the treating physician, no such treatment is available or indicated
* Performance status 0-2 (Per Eastern Cooperative Oncology Group (ECOG) criteria)
* Patients must have acceptable organ function as defined below. However, as noted above, drug-specific inclusion/exclusion criteria specified in the protocol appendix for each agent will take precedence for this and all inclusion criteria:

  1. Absolute neutrophil count ≥ 1.5 x 106/µl
  2. Hemoglobin > 9.0 g/dl
  3. Platelets > 75,000/µl
  4. Total bilirubin < 2.0 mg/ dl, except in patients with Gilbert's Syndrome
  5. Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) < 2.5 x institutional upper limit of normal (ULN) (or < 5 x ULN in patients with known hepatic metastases)
  6. Serum creatinine ≤ 1.5 × ULN or calculated or measured creatinine clearance ≥ 50 mL/min/1.73 m2
* Patients must have disease that can be objectively measured by physical or radiographic exam (per RECIST v1.1 for solid tumor, Lugano criteria for non-Hodgkin lymphoma or International Myeloma Working Group criteria for multiple myeloma), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or a subcutaneous or superficial lesion that can be measured with calipers by clinical exam. For lymph nodes, the short axis must be ≥15 mm. Patient's whose disease cannot be objectively measured by physical or radiographic examination (e.g., elevated serum tumor marker only, bone-only disease without an identifiable soft tissue component, or patients with only assessable non-measurable disease) are NOT eligible.
* Results must be available from a genomic test or immunohistochemistry (IHC) test for protein expression performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified and College of American Pathologists (CAP)-accredited or New York State accredited (for labs offering services to residents of NY) laboratory. Labs that have registered the test with the NIH Genetic Testing Registry or that provide a report that has been designated as optimized for TAPUR participation are preferred, but not required. The genomic or IHC test used to qualify a patient for participation in TAPUR may have been performed on any specimen of the patient's tumor obtained at any point during the patient's care at the discretion of the patient's treating physician. Genomic assays performed on cell-free DNA in plasma ("liquid biopsies") will also be acceptable if the genomic analysis is performed in a laboratory that meets the criteria described above.
* Ability to understand and the willingness to sign a written informed consent/assent document.
* Have a tumor genomic profile for which single agent treatment with one of the FDA approved targeted anti-cancer drugs included in this study has potential clinical benefit based on the criteria described in protocol.
* For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
* Because of the risks of drug treatment to the developing fetus, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for four months following completion of study therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study or if she is the partner of a male participant in this study and becomes pregnant while he is participating in this study, she should inform her or her partner's treating physician immediately as well as her obstetrician. Female study patients who become pregnant must immediately discontinue treatment with any study therapy. Male patients should avoid impregnating a female partner. Male study patients, even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and for a specified amount of time the last dose of study drug, or completely abstain from sexual intercourse.

Note: TAPUR does not explicitly exclude any type of solid tumor, but the patient must have measurable and evaluable disease per RECIST v1.1.

Exclusion Criteria:

* Patients whose disease is not measurable or cannot be assessed by radiographic imaging or physical examination (e.g., elevated serum tumor marker only) are not eligible
* Patients with primary brain tumors or leptomeningeal metastases are excluded.
* Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within the 3 months prior to registration. All patients with previously treated brain metastases must be clinically stable for at least 1 month after completion of treatment and off steroid treatment for one month prior to study enrollment.
* Patients with known progressive brain metastases are eligible but additional eligibility criteria apply.

Note: there are additional exclusion criteria that may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2016-03-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate defined as % of participants in a cohort with complete or partial response or with stable disease according to standard response criteria | Assessed at 16 weeks of treatment
  Each cohort includes participants with the same tumor type, genomic variant and study drug. For solid tumors, the Response Evaluation Criteria for Solid Tumors (RECIST) criteria will be used, for non-Hodgkin Lymphoma, the Lugano Criteria will be used, and for multiple myeloma, the International Uniform Response Criteria for Multiple Myeloma will be used.

SECONDARY OUTCOMES:
Overall survival (OS) | Duration of survival from registration on study until death from any cause, assessed throughout end of study, up to 3 years
  OS will be estimated using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Locations (156):
- United States (156):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Cancer Treatment Centers of America-Phoenix, Phoenix, Arizona
  - Sutter Auburn, Auburn, California
  - Sutter Alta Bates, Berkeley, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - Kaiser Permanente - Oakland Medical Center, Oakland, California
  - Sutter Palo Alto Medical Foundation: Palo Alto, Palo Alto, California
  - Kaiser Permanente - Roseville Medical Center, Roseville, California
  - Sutter Roseville, Roseville, California
  - Kaiser Permanente - Sacramento Medical Center, Sacramento, California
  - Sutter Sacramento, Sacramento, California
  - Kaiser Permanente - South San Francisco Medical Center, San Francisco, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - Sutter Cancer Research Consortium, San Francisco, California
  - Kaiser Permanente - San Jose Medical Center, San Jose, California
  - Kaiser Permanente - San Leandro Medical Center, San Leandro, California
  - Kaiser Permanente - Santa Clara Medical Center, Santa Clara, California
  - Sutter Palo Alto Medical Foundation: Santa Cruz, Santa Cruz, California
  - Sutter Palo Alto Medical Foundation: Fremont, Santa Cruz, California
  - Sutter Palo Alto Medical Foundation: Sunnyvale, Sunnyvale, California
  - Kaiser Permanente - Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente - Walnut Creek Medical Center, Walnut Creek, California
  - Saint Vincent's Medical Center (SVMC), Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center (MSMC), Meriden, Connecticut
  - The Hospital of Central Connecticut (HOCC) Cancer Center, New Britain, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - Charlotte Hungerford, Torrington, Connecticut
  - Windham Hospital (WH), Willimantic, Connecticut
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Altamonte Springs, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Bonita Springs, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Bradenton, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Brandon, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Cape Coral, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Fort Myers, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Gainesville, Florida
  - University of Florida Health, Gainesville, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Largo, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Lecanto, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Naples, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Ocala, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Orange City, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Orlando, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Port Charlotte, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Sarasota, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Tampa, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Tavares, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, The Villages, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Trinity, Florida
  - Florida Cancer Specialists South / Sarah Cannon Research Institute, Venice, Florida
  - Florida Cancer Specialists North / Sarah Cannon Research Institute, Winter Park, Florida
  - Cancer Treatment Centers of America - Atlanta, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Gynecologic Oncology and Surgical Specialists at the Lewis Cancer & Research Pavilion, Savannah, Georgia
  - Lewis Cancer & Research Pavilion at the Melanoma, Skin Cancer & Sarcoma Institute, Savannah, Georgia
  - Lewis Cancer & Research Pavilion, Savannah, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - The Queen's Medical Center - POB I, Honolulu, Hawaii
  - The Queen's Medical Center - Punchbowl, Honolulu, Hawaii
  - The Queen's Medical Center - Kuakini, Honolulu, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Cancer Treatment Centers of America-Chicago, Chicago, Illinois
  - Community Health Network (The University of Texas MD Anderson Cancer Center), Indianapolis, Indiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Jackson Laboratory - Maine Cancer Genomics Initiative, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - SMHC Cancer Care and Blood Disorders -Biddeford, Biddeford, Maine
  - Northern Light Cancer Care, Brewer, Maine
  - Raish Peavey Haskell Children's Cancer and Treatment Center, Brewer, Maine
  - MaineHealth Cancer Care -Brunswick, Brunswick, Maine
  - New England Cancer Specialist, Kennebunk, Maine
  - York Hopsital Oncology & Infusion Care in Kittery, Kittery, Maine
  - Stephens Memorial Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - SMHC Cancer Care and Blood Disorders -Sandford, Sanford, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Maine Medical Partner's Women's Health, Scarborough, Maine
  - New England Cancer Specialist, Scarborough, Maine
  - MaineHealth Cancer Care -South Portland, South Portland, Maine
  - New England Cancer Specialist, Topsham, Maine
  - York Hospital Oncology & Infusion Care in Wells, Wells, Maine
  - York Hospital Oncology & Infusion Care in York, York Village, Maine
  - Trinity Health Ann Arbor Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Livonia Hospital, Livonia, Michigan
  - Trinity Health Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Michigan Cancer Research Consortium, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NH Oncology - Hematology, PA, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - New England Cancer Specialist, Portsmouth, New Hampshire
  - Lovelace Medical Center - Saint Joseph Square, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - The University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center, Rio Rancho, New Mexico
  - Northwell Health Monter Cancer Center, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye, Ear, and Throat Hospital, New York, New York
  - Staten Island University Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Phelps Hospital, Sleepy Hollow, New York
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Atrium Health's Levine Cancer Institute, Charlotte, North Carolina
  - Sanford Health- Bismarck, Bismarck, North Dakota
  - Sanford Health- Fargo, Fargo, North Dakota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Kettering Health, Kettering, Ohio
  - West Chester Hospital, West Chester, Ohio
  - Providence Health & Services, Portland, Oregon
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital- Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - SC Cancer Specialists at St. Joseph's/Candler Bluffton, Bluffton, South Carolina
  - St. Joseph's/Candler Smith, Bluffton, South Carolina
  - Summit Cancer Care at St. Josph's/Candler Bluffton, Bluffton, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Sanford Cancer Center Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - Tennessee Oncology - Nashville / Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cedar City Hospital, SW Cancer Clinic, Sandra Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - Dixie Regional Medical Center-River Road Campus, St. George, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Aurora Cancer Care - Burlington, Burlington, Wisconsin
  - Aurora Health Care - Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care - Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care - Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Cancer Care Milwaukee, Milwaukee, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Aurora West Allis Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care - Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Center, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care - Milwaukee West, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Carrizosa DR, Rothe M, Mangat PK, Garrett-Mayer E, Behl D, Adesunloye B, Pisick E, Beekman KW, Dotan E, Akce M, Alese OB, Sahai V, Klute KA, Aragon-Ching JB, Cooper KA, Thota R, Meric-Bernstam F, Hosein PJ, Maestas EC, Moyers JT, Powell S, Zhao S, Hobbs E, Rueter J, Sohal DPS, Taylor MA, Hinshaw DC, Gregory A, Grantham GN, Halabi S, Schilsky RL. Olaparib in Patients With Solid Tumors With ATM Alterations: Results From the Targeted Agent and Profiling Utilization Registry (TAPUR) Study. JCO Precis Oncol. 2026 Jan;10:e2500716. doi: 10.1200/PO-25-00716. Epub 2026 Jan 15. PMID 41538762
- [Derived] Al Baghdadi T, Rothe M, Mangat PK, Garrett-Mayer E, Crysler OV, Mileham KF, Farrington LC, Adesunloye B, Dublis SA, Astsaturov I, Calfa CJ, Bleeker J, Khalil M, Thota R, Cannon TL, Alese OB, Gold PJ, Hafez N, Baron AD, Meric-Bernstam F, Hobbs E, Marr AS, Rueter J, Tawfik B, Hinshaw DC, Gregory A, Grantham GN, Halabi S, Schilsky RL. Olaparib in Patients With Solid Tumors With BRCA1/2 Alterations: Results From The Targeted Agent and Profiling Utilization Registry (TAPUR) Study. JCO Precis Oncol. 2025 Oct;9:e2500649. doi: 10.1200/PO-25-00649. Epub 2025 Oct 16. PMID 41100773
- [Derived] Mangat PK, Kirkwood MK, Hinshaw DC, Garrett-Mayer E, Schilsky RL. Prevalence of targetable genomic alterations among a diverse population participating in the ASCO TAPUR Study. NPJ Precis Oncol. 2025 Jul 3;9(1):222. doi: 10.1038/s41698-025-00962-1. PMID 40610648
- [Derived] Worden FP, Pisick E, Rothe M, Mangat PK, Garrett-Mayer E, Khalil MF, Carrizosa DR, Bauman JR, Leidner RS, Duvivier HL, Fu S, Park MS, Yost KJ, Calfa CJ, Marr AS, Balmanoukian AS, Behl D, Cannon TL, Nabell L, Powell SF, Thota R, Hinshaw DC, Gregory A, Grantham GN, Halabi S, Schilsky RL. Palbociclib in Patients With Head and Neck Cancer and Other Tumors With CDKN2A Alterations: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2024 Oct;8:e2400477. doi: 10.1200/PO-24-00477. Epub 2024 Oct 16. PMID 39413339
- [Derived] Schuetze S, Rothe M, Mangat PK, Garrett-Mayer E, Meric-Bernstam F, Calfa CJ, Farrington LC, Livingston MB, Wentzel K, Behl D, Kier Y, Marr AS, von Mehren M, Press JZ, Thota R, Grantham GN, Gregory A, Hinshaw DC, Halabi S, Schilsky RL. Palbociclib in Patients With Soft Tissue Sarcoma With CDK4 Amplifications: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2024 Jul;8:e2400219. doi: 10.1200/PO.24.00219. PMID 39013131
- [Derived] Srkalovic G, Rothe M, Mangat PK, Garrett-Mayer E, Ahn ER, Brouse G, Chan J, Mehmi I, Khalil M, Duvivier HL, Gaba A, Leuva H, Thota R, Yost KJ, Grantham GN, Gregory A, Hinshaw DC, Halabi S, Schilsky RL. Talazoparib in Patients With Solid Tumors With BRCA1/2 Mutation: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2024 Jun;8:e2400026. doi: 10.1200/PO.24.00026. PMID 38865672
- [Derived] Cannon TL, Rothe M, Mangat PK, Garrett-Mayer E, Chiu VK, Hwang J, Vijayvergia N, Alese OB, Dib EG, Duvivier HL, Klute KA, Sahai V, Ahn ER, Bedano P, Behl D, Sinclair S, Thota R, Urba WJ, Yang ES, Grantham GN, Hinshaw DC, Gregory A, Halabi S, Schilsky RL. Pertuzumab Plus Trastuzumab in Patients With Biliary Tract Cancer With ERBB2/3 Alterations: Results From the Targeted Agent and Profiling Utilization Registry Study. J Clin Oncol. 2024 Sep 20;42(27):3228-3237. doi: 10.1200/JCO.23.02078. Epub 2024 May 15. PMID 38748939
- [Derived] Perez JK, Kleber J, Rothe M, Mangat P, Garrett-Mayer E, Schilsky RL. Concordance in Molecular Tumor Board Case Reviews in the ASCO TAPUR Study. JCO Precis Oncol. 2024 Mar;8:e2300615. doi: 10.1200/PO.23.00615. PMID 38564684
- [Derived] Calfa CJ, Rothe M, Mangat PK, Garrett-Mayer E, Ahn ER, Burness ML, Gogineni K, Rohatgi N, Al Baghdadi T, Conlin A, Gaba A, Hamid O, Krishnamurthy J, Gavini NJ, Gold PJ, Rodon J, Rueter J, Thota R, Grantham GN, Hinshaw DC, Gregory A, Halabi S, Schilsky RL. Sunitinib in Patients With Breast Cancer With FGFR1 or FGFR2 Amplifications or Mutations: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2024 Feb;8:e2300513. doi: 10.1200/PO.23.00513. PMID 38354330
- [Derived] Meric-Bernstam F, Rothe M, Mangat PK, Garrett-Mayer E, Gutierrez R, Ahn ER, Cannon TL, Powell S, Krauss JC, Reynolds CM, von Mehren M, Behl D, Calfa CJ, Duvivier HL, Kaplan HG, Livingston MB, Sharma MR, Urba WJ, Grantham GN, Hinshaw DC, Gregory A, Halabi S, Schilsky RL. Cobimetinib Plus Vemurafenib in Patients With Solid Tumors With BRAF Mutations: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2023 Sep;7:e2300385. doi: 10.1200/PO.23.00385. PMID 38096472
- [Derived] Rohatgi N, Rothe M, Mangat PK, Garrett-Mayer E, Meric-Bernstam F, Pisick E, Alese OB, Reynolds CM, Thota R, Vaccaro GM, von Mehren M, Arend RC, Chiu VK, Duvivier HL, Gold PJ, Hack K, Marr AS, Winer A, Grantham GN, Hinshaw DC, Gregory A, Halabi S, Schilsky RL. Nivolumab Plus Ipilimumab in Patients With Solid Tumors With ATM Mutations: Results From the Targeted Agent and Profiling Utilization Registry (TAPUR) Study. JCO Precis Oncol. 2023 Sep;7:e2300279. doi: 10.1200/PO.23.00279. PMID 38039429
- [Derived] Duvivier HL, Rothe M, Mangat PK, Garrett-Mayer E, Ahn ER, Al Baghdadi T, Alva AS, Dublis SA, Cannon TL, Calfa CJ, Li R, Behl D, Chiu VK, Gold PJ, Marr AS, Mileham KF, Powell SF, Rodon J, Thota R, Grantham GN, Gregory A, Hinshaw DC, Halabi S, Schilsky RL. Pembrolizumab in Patients With Tumors With High Tumor Mutational Burden: Results From the Targeted Agent and Profiling Utilization Registry Study. J Clin Oncol. 2023 Nov 20;41(33):5140-5150. doi: 10.1200/JCO.23.00702. Epub 2023 Aug 10. PMID 37561967
- [Derived] Mangat PK, Garrett-Mayer E, Perez JK, Schilsky RL. The Targeted Agent and Profiling Utilization Registry Study: A pragmatic clinical trial. Clin Trials. 2023 Dec;20(6):699-707. doi: 10.1177/17407745231182013. Epub 2023 Jul 25. PMID 37489819
- [Derived] Ganti AK, Rothe M, Mangat PK, Garrett-Mayer E, Dib EG, Duvivier HL, Ahn ER, Behl D, Borghaei H, Balmanoukian AS, Gaba A, Li R, Osei-Boateng K, Thota R, Grantham GN, Gregory A, Halabi S, Schilsky RL. Pertuzumab Plus Trastuzumab in Patients With Lung Cancer With ERBB2 Mutation or Amplification: Results From the Targeted Agent and Profiling Utilization Registry Study. JCO Precis Oncol. 2023 Jun;7:e2300041. doi: 10.1200/PO.23.00041. PMID 37315265
- [Derived] Ahn ER, Rothe M, Mangat PK, Garrett-Mayer E, Ali-Ahmad HM, Chan J, Maitland ML, Patel SR, Reese Z, Balmanoukian AS, Drescher CW, Li R, Tsimberidou AM, Leath CA 3rd, O'Lone R, Grantham GN, Halabi S, Schilsky RL. Pertuzumab Plus Trastuzumab in Patients With Endometrial Cancer With ERBB2/3 Amplification, Overexpression, or Mutation: Results From the TAPUR Study. JCO Precis Oncol. 2023 Apr;7:e2200609. doi: 10.1200/PO.22.00609. PMID 37027810
- [Derived] Yang ES, Halabi S, Rothe M, Garrett-Mayer E, Mangat PK, Pisick E, Dib E, Burgess EF, Zakem M, Rohatgi N, Bilen MA, O'Lone R, Grantham GN, Schilsky RL. Olaparib in Patients With Metastatic Prostate Cancer With BRCA1/2 Mutation: Results From the TAPUR Study. JCO Precis Oncol. 2023 Feb;7:e2200505. doi: 10.1200/PO.22.00505. PMID 36753688
- [Derived] Gupta R, Meric-Bernstam F, Rothe M, Garrett-Mayer E, Mangat PK, D'Andre S, Ahn ER, O'Lone R, Halabi S, Grantham GN, Schilsky RL. Pertuzumab Plus Trastuzumab in Patients With Colorectal Cancer With ERBB2 Amplification or ERBB2/3 Mutations: Results From the TAPUR Study. JCO Precis Oncol. 2022 Oct;6:e2200306. doi: 10.1200/PO.22.00306. PMID 36315917
- [Derived] Alva AS, Mangat PK, Garrett-Mayer E, Halabi S, Hansra D, Calfa CJ, Khalil MF, Ahn ER, Cannon TL, Crilley P, Fisher JG, Haslem DS, Shrestha S, Antonelli KR, Butler NL, Warren SL, Rygiel AL, Ranasinghe S, Bruinooge SS, Schilsky RL. Pembrolizumab in Patients With Metastatic Breast Cancer With High Tumor Mutational Burden: Results From the Targeted Agent and Profiling Utilization Registry (TAPUR) Study. J Clin Oncol. 2021 Aug 1;39(22):2443-2451. doi: 10.1200/JCO.20.02923. Epub 2021 Apr 12. PMID 33844595
- [Derived] Fisher JG, Tait D, Garrett-Mayer E, Halabi S, Mangat PK, Schink JC, Alvarez RH, Veljovich D, Cannon TL, Crilley PA, Pollock T, Calfa CJ, Al Baghdadi T, Thota R, Fleming N, Cotta JA, Rygiel AL, Warren SL, Schilsky RL. Cetuximab in Patients with Breast Cancer, Non-Small Cell Lung Cancer, and Ovarian Cancer Without KRAS, NRAS, or BRAF Mutations: Results from the Targeted Agent and Profiling Utilization Registry (TAPUR) Study. Target Oncol. 2020 Dec;15(6):733-741. doi: 10.1007/s11523-020-00753-7. PMID 33090333
- [Derived] Al Baghdadi T, Garrett-Mayer E, Halabi S, Mangat PK, Rich P, Ahn ER, Chai S, Rygiel AL, Osayameh O, Antonelli KR, Islam S, Bruinooge SS, Schilsky RL. Sunitinib in Patients with Metastatic Colorectal Cancer (mCRC) with FLT-3 Amplification: Results from the Targeted Agent and Profiling Utilization Registry (TAPUR) Study. Target Oncol. 2020 Dec;15(6):743-750. doi: 10.1007/s11523-020-00752-8. PMID 33068284